CLINICAL TRIAL: NCT07389564
Title: NOVEL-HF - Nationwide Registry of Patients With Heart Failure With Improved and Supranormal Ejection Fraction
Brief Title: Nationwide Registry of Patients With Heart Failure With Improved and Supranormal Ejection Fraction
Acronym: NOVEL-HF
Status: Active, not recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Konrad Stępień, MD, PhD, Jagiellonian University
Other Study IDs: 86/KBL/OIL/2025
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: heart failure; registry; prognosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure with improved ejection fraction: Patients with HF with an initial left ventricular ejection fraction (LVEF) below 40%, with at least a 10% increase during follow-up, and with final values >40%
- Heart failure with supranormal ejection fraction: Patients with HF whose LVEF values on echocardiography are >65%

SUMMARY:
NOVEL-HF is a multicenter, observational nationwide registry of HFimpEF and HFsnEF conducted in cooperation with the Scientific Platform of the Polish Society of Cardiology.

According to the current definitions the criteria for HFimpEF diagnosis include patients with HF with an initial left ventricular ejection fraction (LVEF) below 40%, with at least a 10% increase during follow-up, and with final values >40%. HFsnEF includes patients with HF whose LVEF values on echocardiography are >65%.

The patient data will be collected from standardized and anonymous forms via the Scientific Platform of the Polish Society of Cardiology. The NOVEL-HF registry will involve the complete clinical, laboratory, and echocardiographic characteristics, as well as introduced pharmacological treatment. The occurrence of end-points (all-cause mortality, cardiovascular mortality, HF decompensations, worsening of HF symptoms) will be assessed in short- and long-term follow-up.

In accordance with initial assumptions, 500 HFimpEF and 200 HFsnEF patients in all participating centers will be included.

Ethical approval was granted by the local Bioethics Committee.

DETAILED DESCRIPTION:
Heart failure with improved ejection fraction (HFimpEF) and heart failure with supranormal ejection fraction (HFsnEF) are new and poorly understood subtypes of heart failure with significant prognostic implications.

The primary goal of the proposed "Nationwide registry of patients with heart failure with improved and supranormal ejection fraction (NOVEL-HF)" is to comprehensively characterize the Polish population of patients with HFimpEF and HFsnEF.

The collected data will allow for understanding their etiology, determining detailed clinical characteristics, and predictors of mortality in both short and long-term follow-up. Once a sufficient number of patients are enrolled, new prognostic scoring scales will be developed based on NOVEL-HF registry data to aid in predicting prognosis in these patient groups.

Each participating center will enroll patients > 18 years old retrospectively from their internal databases based on the clinical and echocardiographic diagnosis of HFimpEF and HFsnEF, but also prospectively for six months from the NOVEL-HF joining with informed consent of the patients.

NOVEL-HF is a multicenter, observational nationwide registry of HFimpEF and HFsnEF conducted in cooperation with the Scientific Platform of the Polish Society of Cardiology.

According to the current definitions the criteria for HFimpEF diagnosis include patients with HF with an initial left ventricular ejection fraction (LVEF) below 40%, with at least a 10% increase during follow-up, and with final values >40% [1]. HFsnEF includes patients with HF whose LVEF values on echocardiography are >65%.

The patient data will be collected from standardized and anonymous forms via the Scientific Platform of the Polish Society of Cardiology. The NOVEL-HF registry will involve the complete clinical, laboratory, and echocardiographic characteristics, as well as introduced pharmacological treatment. The occurrence of end-points (all-cause mortality, cardiovascular mortality, HF decompensations, worsening of HF symptoms) will be assessed in short- and long-term follow-up.

In accordance with initial assumptions, 500 HFimpEF and 200 HFsnEF patients in all participating centers will be included.

Ethical approval was granted by the local Bioethics Committee.

Data obtained from the NOVEL-HF registry will enable understanding the HFimpEF and HFsnEF etiology, determining detailed clinical characteristics, and predictors of mortality in both short and long-term follow-up. Once a sufficient number of patients are enrolled, new prognostic scoring scales will be developed based on NOVEL-HF registry data to aid in predicting prognosis in these patient groups.

It was planned to prepare at least 5 full-text publications in peer-reviewed Polish (Polish Heart Journal) and foreign journals.

The condition for participation in NOVEL-HF and the planned publications is the inclusion of at least 50 patients with HFimpEF and/or 20 patients with HFsnEF.

ELIGIBILITY:
Inclusion Criteria:

* HFimpEF or HFsnEF diagnosis

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each participating center will enroll patients > 18 years old retrospectively from their internal databases based on the clinical and echocardiographic diagnosis of HFimpEF and HFsnEF, but also prospectively for six months from the NOVEL-HF joining with informed consent of the patients.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months
  All-cause mortality

SECONDARY OUTCOMES:
Cardiovascular mortality | 12 months
  Cardiovascular mortality
HF decompensations | 12 months
  HF decompensations
Worsening of HF symptoms | 12 months
  Worsening of HF symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Coronary Disease and Heart Failure, John Paul II Hospital in Krakow, Jagiellonian University Medical College, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stepien K, Eliasz K, Nowak K, Karcinska A, Kachnic N, Yika ADC, Platschek M, Krawczyk K, Siniarski A, Zalewski J, Nessler J. Clinical determinants and long-term survival in heart failure with supra-normal ejection fraction. Insights from LECRA-HF registry. Adv Med Sci. 2025 Mar;70(1):166-171. doi: 10.1016/j.advms.2025.02.005. Epub 2025 Feb 19. PMID 39983867
- [Result] Stepien K, Nowak K, Kachnic N, Karcinska A, Del Carmen Yika A, Furczynski J, Platschek M, Skorupa M, Wylecial Z, Zalewski J, Nessler J. Clinical characteristics and long-term outcomes of patients with heart failure with improved ejection fraction. First Polish experience from LECRA-HF registry. Adv Med Sci. 2024 Mar;69(1):132-138. doi: 10.1016/j.advms.2024.02.009. Epub 2024 Mar 4. PMID 38447613